CLINICAL TRIAL: NCT03880578
Title: Influence of Radioiodine Treatment on Thyroid Function and Quality of Life of Patients
Brief Title: Quality of Life After Interventional Thyroid Treatment
Acronym: DSR
Status: Completed | Type: Observational
Sponsor: Klinikum Lüdenscheid (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01-30/R3; 2019-01-30/R3 (Other: Klinikum Luedenscheid)
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-01

CONDITIONS: Thyroid; Deficiency; Quality of Life
Keywords: LT4 treatment; QoL
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- surgery (withdrawn, not continuing recruiting): thyroid patients receiving replacement treatment with levothyroxine (LT4) after thyroidectomy
  Interventions: Drug: Levothyroxine Sodium
- radioiodine: thyroid patients receiving replacement treatment with levothyroxine (LT4) following radioiodine treatment
  Interventions: Drug: Levothyroxine Sodium
- control: thyroid patients followed without surgery or radioiodine treatment
  Interventions: Drug: Levothyroxine Sodium

INTERVENTIONS:
Drug: Levothyroxine Sodium — thyroid hormone replacement
  Other Names: LT4

SUMMARY:
In this study, patients are prospectively followed after radioiodine treatment to assess the relationship between thyroid status and their quality of life after thyroid ablative treatment.

A third treatment arm after surgery has been stopped, as deemed currently not feasible to achieve its target.

DETAILED DESCRIPTION:
Patients are frequently dissatisfied with LT4 replacement treatment. The reasons for persisting patient complaints are poorly understood. Conversion efficiency and impaired T3/T4 ratios in athyreotic patients may play a major role. We hypothesised that the extent of ablation either by surgery or radioiodine treatment may result in biochemical disequilibria between FT3, FT4 and TSH and those may be, in turn, associated with persisting symptomatology.

The study follows patients after radioiodine therapy as well as a control group over half a year, assessing thyroid status, set points, conversion rates, thyroid volume, LT4 administration and dosing, demographic characteristics and quality of life measures. The treatment mode is not part of the study, and determined by criteria and procedures of best standard care. For that reason, a randomised or blinded design is not possible.

Changes and interrelationships between thyroid parameters and QoL measures are analysed within-subjects and between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a thyroid disease requiring radioiodine treatment
* Clinical diagnosis of a thyroid disease requiring follow-up but no ablative treatment (controls)
* Clinical diagnosis of a thyroid disease requiring surgery stopped recruiting

Exclusion Criteria:

* paediatric patients
* interfering comorbidity
* non-thyroidal illness
* pregnancy
* psychiatric disease
* severe psychological disorder
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: thyroid patients in a routine ambulatory setting specialising in Nuclear Medicine
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Larisch, Professor, Principal Investigator — Director of Department; Rudolf Hoermann, Professor, Study Chair — Klinikum Lüdenscheid
Locations (1):
- Department of Nuclear Medicine Klinikum Luedenscheid, Lüdenscheid, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data are principally shared depending on compliance with relevant regulations and authorisation

REFERENCES:
- [Background] Larisch R, Midgley JEM, Dietrich JW, Hoermann R. Symptomatic Relief is Related to Serum Free Triiodothyronine Concentrations during Follow-up in Levothyroxine-Treated Patients with Differentiated Thyroid Cancer. Exp Clin Endocrinol Diabetes. 2018 Sep;126(9):546-552. doi: 10.1055/s-0043-125064. Epub 2018 Feb 2. PMID 29396968
- [Background] Hoermann R, Midgley JEM, Larisch R, Dietrich JW. Recent Advances in Thyroid Hormone Regulation: Toward a New Paradigm for Optimal Diagnosis and Treatment. Front Endocrinol (Lausanne). 2017 Dec 22;8:364. doi: 10.3389/fendo.2017.00364. eCollection 2017. PMID 29375474
- [Background] Hoermann R, Midgley JEM, Larisch R, Dietrich JW. The role of functional thyroid capacity in pituitary thyroid feedback regulation. Eur J Clin Invest. 2018 Oct;48(10):e13003. doi: 10.1111/eci.13003. Epub 2018 Aug 1. PMID 30022470
- [Background] Hoermann R, Midgley JE, Larisch R, Dietrich JW. Homeostatic Control of the Thyroid-Pituitary Axis: Perspectives for Diagnosis and Treatment. Front Endocrinol (Lausanne). 2015 Nov 20;6:177. doi: 10.3389/fendo.2015.00177. eCollection 2015. PMID 26635726
- [Background] Hoermann R, Midgley JEM, Larisch R, Dietrich JWC. Advances in applied homeostatic modelling of the relationship between thyrotropin and free thyroxine. PLoS One. 2017 Nov 20;12(11):e0187232. doi: 10.1371/journal.pone.0187232. eCollection 2017. PMID 29155897
- [Background] Midgley JE, Larisch R, Dietrich JW, Hoermann R. Variation in the biochemical response to l-thyroxine therapy and relationship with peripheral thyroid hormone conversion efficiency. Endocr Connect. 2015 Dec;4(4):196-205. doi: 10.1530/ec-150056. PMID 26335522
- [Background] Hoermann R, Midgley JE, Larisch R, Dietrich JW. Is pituitary TSH an adequate measure of thyroid hormone-controlled homoeostasis during thyroxine treatment? Eur J Endocrinol. 2013 Jan 17;168(2):271-80. doi: 10.1530/EJE-12-0819. Print 2013 Feb. PMID 23184912
- [Background] Winther KH, Cramon P, Watt T, Bjorner JB, Ekholm O, Feldt-Rasmussen U, Groenvold M, Rasmussen AK, Hegedus L, Bonnema SJ. Disease-Specific as Well as Generic Quality of Life Is Widely Impacted in Autoimmune Hypothyroidism and Improves during the First Six Months of Levothyroxine Therapy. PLoS One. 2016 Jun 3;11(6):e0156925. doi: 10.1371/journal.pone.0156925. eCollection 2016. PMID 27257805
- [Background] Dietrich JW, Landgrafe-Mende G, Wiora E, Chatzitomaris A, Klein HH, Midgley JE, Hoermann R. Calculated Parameters of Thyroid Homeostasis: Emerging Tools for Differential Diagnosis and Clinical Research. Front Endocrinol (Lausanne). 2016 Jun 9;7:57. doi: 10.3389/fendo.2016.00057. eCollection 2016. PMID 27375554

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery (Withdrawn, Not Continuing Recruiting) | Radioiodine | Control
Started | 0 | 51 | 50
12 Months | 0 | 14 | 19
Completed | 0 | 47 | 49
Not Completed | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: euthyroid patients presenting at fixed intervals for surveillance of non-toxic nodular goitre
- Radioiodine: Untreated patients with subclinical hyperthyroidism referred for radioiodine treatment
- Total: Total of all reporting groups
Arm/Group | Control | Radioiodine | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (14.1) | 61.6 (12.5) | 55.4 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 50 | 51 | 101
Region of Enrollment [Number; unit: participants]
  Germany | 50 | 51 | 101
FT3 [Mean (Standard Deviation); unit: pmol/L] | 5.32 (0.70) | 5.45 (0.71) | 5.39 (0.70)
FT4 [Mean (Standard Deviation); unit: pmol/L] | 15.4 (2.02) | 15.3 (2.29) | 15.3 (2.15)
TSH [Median (Inter-Quartile Range); unit: mIU/L] | 1.25 [0.91 to 1.79] | 0.39 [0.24 to 0.56] | 0.75 [0.39 to 1.26]
Thyroid volume [Mean (Standard Deviation); unit: ml] | 19.8 (10.3) | 29.7 (14.2) | 24.7 (13.3)

OUTCOME MEASURES:

1. Primary Outcome: ThyPRO Scale Scores (0-100, Higher Scores Indicating Worse Quality of Life)
Description: quality of life measured by a thyroid specific validated questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score
Groups:
- Control; Radioiodine: Composite ThyPRO score
Arm/Group | Control | Radioiodine
Number analyzed (Participants) | 50 | 51
score | 18.3 (10.8) | 19.9 (14.8)
Statistical Analysis 1: Comparison: Control vs Radioiodine; Test type: Superiority; p < 0.001, Mixed Models Analysis; The outcome measure is change over time between treatment groups, reported as a mean adjusted difference; Mean Difference (Final Values) = -10.3, 95% CI 2-sided [-14.9 to -5.7] — change in the composite score of the ThyPRO between groups

2. Secondary Outcome: Rate of Global Deiodinase Activity (SPINA-GD, See Reference Calculated Parameters)
Description: efficiency of converting T4 into T3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: nmol/s
Groups:
- Control: Control group
- Radioiodine: Treatment group
Arm/Group | Control | Radioiodine
Number analyzed (Participants) | 50 | 51
nmol/s | 32.9 (5.03) | 32.2 (5.52)
Statistical Analysis 1: Comparison: Control vs Radioiodine; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-4.34 to 0.06]

3. Other Pre Specified Outcome: Serum Concentration of TSH
Description: TSH
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mIU/L
Groups:
- Control; Radioiodine: TSH
Arm/Group | Control | Radioiodine
Number analyzed (Participants) | 50 | 51
mIU/L | 1.39 (0.63) | 2.34 (2.58)
Statistical Analysis 1: Comparison: Control vs Radioiodine; Test type: Superiority; p < 0.001, Mixed Models Analysis; Median Difference (Final Values) = 1.70, 95% CI 2-sided [1.27 to 2.03] — MAD obtained after log transformation of TSH

4. Other Pre Specified Outcome: Serum Concentrations of FT3 and FT4
Description: Thyroid hormones FT3, FT4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Control; Radioiodine: Thyroid hormones FT3, FT4
Arm/Group | Control | Radioiodine
Number analyzed (Participants) | 50 | 51
pmol/L
  FT3 | 5.33 (0.60) | 4.84 (0.65)
  FT4 | 15.2 (2.13) | 14.2 (2.38)
Statistical Analysis 1: Comparison: Control vs Radioiodine; FT3; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.87 to -0.35]
Statistical Analysis 2: Comparison: Control vs Radioiodine; FT4; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.81 to 0.15]

5. Other Pre Specified Outcome: Thyroid Volume Measured by Ultrasound (ml)
Description: thyroid capacity
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Control | Radioiodine
Number analyzed (Participants) | 50 | 51
ml | 20.5 (12.8) | 18.8 (10.3)
Statistical Analysis 1: Comparison: Control vs Radioiodine; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-14.6 to -8.5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Radioiodine
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT03880578/Prot_SAP_000.pdf